CLINICAL TRIAL: NCT01954628
Title: The FLAGSHIP Study: A 12-week Phase II Study to Evaluate the Efficacy and Safety of AQX-1125 Following Exacerbations in Patients With Chronic Obstructive Pulmonary Disease (COPD) by Targeting the SHIP1 Pathway
Brief Title: Efficacy and Safety of AQX-1125 in Unstable COPD
Acronym: FLAGSHIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aquinox Pharmaceuticals (Canada) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AQX-1125-202
Record Dates: First submitted 2013-09-21; First posted 2013-10-07 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: COPD
Keywords: Exacerbation of COPD; Unstable COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — 4-(4-(aminomethyl)-7a-methyl-1-methylideneoctahydro-1H-inden-5-yl)-3-(hydroxymethyl)-4-methylcyclohexan-1-ol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AQX-1125 (Experimental): 1 x AQX-1125 capsule daily
  Interventions: Drug: AQX-1125
- Placebo (Placebo Comparator): 1 x Placebo capsule daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AQX-1125 — Synthetic SHIP1 activator
  Arms: AQX-1125
Drug: Placebo — Placebo control
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effect of 12 weeks of treatment with once daily administration of AQX-1125 compared to placebo in subjects following exacerbations of Chronic Obstructive Pulmonary Disease (COPD) by targeting the SHIP1 (Src Homology 2-containing Inositol-5'-Phosphatase 1) pathway.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a leading cause of morbidity and mortality worldwide. Acute exacerbations of COPD are usually treated with steroids and/or antibiotics. Currently this conventional therapy has significant side effects including osteoporosis, cataracts and suppression of the immune system (from the steroids) and increasing bacterial resistance and other side effects from the use of antibiotics. During an acute exacerbation of COPD, the inflammation in the airways increases.

AQX-1125 represents a new type drug that based current data is thought decrease the inflammatory process and therefore may provide a therapeutic benefit in the treatment of COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥40 years at screening
2. History of COPD for at least 18 months prior to screening, characterised by excessive sputum production
3. Chronic productive cough for at least 3 months in each of the 2 years prior to screening (if other causes of productive cough have been excluded) and/or an exacerbation of COPD with predominantly bronchitic symptoms at enrolment
4. At least 2 documented exacerbations during the last 18 months prior to screening.
5. Presentation of a diagnosed acute exacerbation of COPD, or have recently (within 3 days) been discharged from hospital due to an acute exacerbation of COPD
6. Ability to perform pulmonary function testing and with documented fixed airway obstruction determined by an FEV1 /FVC [forced vital capacity] ratio (post-bronchodilator) of <0.70 and a predicted FEV1 value of 30%-80% of normal within the 6 months prior to Visit 1.
7. Former smoker or current smoker, both with a smoking history of at least 10 pack years

Exclusion Criteria:

1. Diagnosis of other relevant lung disease (e.g. asthma, cystic fibrosis [CF] or significant non-CF bronchiectasis)
2. Known alpha-1-antitrypsin deficiency
3. Treatment with roflumilast or theophylline within 1 month prior to screening
4. Lobar pneumonia, with current positive chest X-ray (CXR) or within the 3 months prior to screening including the presence of any new radiological infiltrate on CXR within the previous two weeks
5. Hospitalisation for more than 7 days for current acute exacerbation, or the requirement for intubation during hospitalisation
6. For outpatients, prior medical history indicating that previous exacerbations required >3 weeks to stabilise

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Shrewsbury, MD, Study Director — Aquinox Pharmaceuticals (Canada) Inc.
Locations (8):
- University of Cincinnati, Cincinnati, Ohio, United States
- Department of Respiratory & Sleep Medicine, Westmead Hospital, Wentworthville, New South Wales, Australia
- Department of Respiratory Medicine, Odense University Hospital, Odense, Denmark
- Biomedicum Helsinki, Helsinki, Finland
- Csongrád Megyei Melkasi Betegségek Szakkórháza, Deszk, Hungary
- P3 Research, Wellington, New Zealand
- Medical University of Lodz, Lodz, Poland
- Lung and Allergy Clinic, Skåne University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GOLD COPD Guidelines — http://goldcopd.org/global-strategy-diagnosis-management-prevention-copd-2016/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 8 countries: Australia, Denmark, Finland, Hungary, New Zealand, Poland, Sweden and US. US subjects participating in 6 month safety follow-up continued in the study until November 2015.
Pre-assignment Details: Four hundred subjects were randomized into two subsets: (1) Subjects suitable for outpatient treatment of a current exacerbation of COPD (within 3 days of diagnosis) & (2) Subjects who had been hospitalized in order to treat their exacerbation for not more than 7 days & were ready to be discharged or had been discharged within the last 3 days.
Groups:
- AQX-1125 (200 mg): AQX-1125 (200 mg capsule), oral once daily for 12 weeks. All standard of care treatments for COPD were permitted throughout the study with the exception of Roflumilast and Theophylline.
- Placebo: Placebo (matching AQX-1125 capsule), oral, once daily for 12 weeks. Placebo control. All standard of care treatments for COPD were permitted throughout the study with the exception of Roflumilast and Theophylline.
Period: Overall Study
Arm/Group | AQX-1125 (200 mg) | Placebo
Started | 200 | 200
Full Analysis Set (FAS) | 200 | 198
Safety Set | 200 | 200
Pharmacokinetic Population | 181 | 0
US 6 Month Ophthalmology Safety Visit | 37 | 32
Completed | 169 | 173
Not Completed | 31 | 27

BASELINE CHARACTERISTICS:
Population: Safety set.
Groups:
- AQX-1125 (200 mg): 1 x AQX-1125 capsule daily
  AQX-1125: Synthetic SHIP1 activator
- Total: Total of all reporting groups
Arm/Group | AQX-1125 (200 mg) | Placebo | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (8.2) | 64.4 (8.5) | 65.1 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 91 | 190
  Male | 101 | 109 | 210
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 193 | 193 | 386
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 9 | 20
  White | 188 | 189 | 377
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 3 | 3 | 6
  Sweden | 0 | 1 | 1
  Hungary | 40 | 43 | 83
  United States | 51 | 53 | 104
  Finland | 5 | 3 | 8
  Denmark | 13 | 13 | 26
  Poland | 81 | 75 | 156
  Australia | 7 | 9 | 16
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 28.1 (6.6) | 27.2 (6.1) | 27.6 (6.3)
Number of COPD Exacerbations in Last 18 months [Mean (Standard Deviation); unit: number of exacerbations/18 months] | 3.1 (1.7) | 3.0 (1.4) | 3.1 (1.5)
Number of Previous Hospitalizations for COPD [Mean (Standard Deviation); unit: number of previous hospitlizations] | 1.1 (3.0) | 0.9 (1.6) | 1.0 (2.4)
Years Since COPD Diagnosis [Mean (Standard Deviation); unit: years] | 8.2 (5.7) | 7.8 (5.9) | 8.0 (5.8)
Smoking Status [Number; unit: participants]
  Current Smokers | 69 | 103 | 172
  Former Smoker | 131 | 97 | 228
Smoking Pack Years [Mean (Standard Deviation); unit: pYears] | 40.2 (22.0) | 41.2 (20.9) | 40.7 (21.4)
Nicotine Replacement Therapy Use [Number; unit: participants]
  Yes | 196 | 195 | 391
  No | 4 | 5 | 9
Post-bronchodilator FEV1/FVC Ratio [Mean (Standard Deviation); unit: ratio] | 0.51 (0.11) | 0.52 (0.11) | 0.52 (0.11)
Post-bronchodilator FEV1% of Predicted [Mean (Standard Deviation); unit: percent predicted] | 50.2 (13.9) | 50.9 (13.2) | 50.6 (13.5)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Variable Was the AAC for Daily EXACT Scores During the 12-week Treatment Period.
Description: The primary variable (endpoint) of this study is the difference in the Area Above the Curve (AAC) for the daily EXACT score from baseline to Week 12 between subjects treated with AQX-1125 and placebo.The EXACT questionnaire is a patient reported outcome (PRO) measure designed to standardise the method for evaluating the frequency, severity and duration of acute exacerbations of COPD. The EXACT is a 14-item daily questionnaire where each item is assessed on a 5 or 6 point ordinal scale. Participants completed the EXACT questionnaire on a daily basis via an electronic diary from Day 1 (pre-dose) to Day 84 (week 12). Higher scores on the daily EXACT questionnaire indicate a more severe health state. When the post-treatment EXACT scores are lower (i.e. improved symptoms) than baseline EXACT, the AACs are positive.
Time Frame: 12 weeks
Population: Full Analysis Set (FAS). The FAS was all randomized subjects who have received at least one dose of the study drug and had at least one efficacy assessment (valid diary entries) post-baseline. Imputation, the mean of the last 5 days, counted backwards from day of last recording, in the treatment period will be used.
Measure: Least Squares Mean (95% Confidence Interval); unit: Area Above Curve on Daily Exact Score
Groups:
- AQX-1125 (200mg): 1 x AQX-1125 capsule daily
Arm/Group | AQX-1125 (200mg) | Placebo
Number analyzed (Participants) | 179 | 183
Area Above Curve on Daily Exact Score | 415.4 [290.7 to 540.1] | 391.7 [268.2 to 515.1]
Statistical Analysis 1: Comparison: AQX-1125 (200mg) vs Placebo; Sample size based on area above the daily EXACT score curve (AAC) from Day 1 to Day 29 from subjects with an acute COPD exacerbation, collected over 28 days. Assuming a residual SD of 500 points, a sample size of 200 subjects per arm would be expected to have an 80% power to detect a true treatment difference in the AAC of 140 points over 12-weeks treatment, using a 2-sided test; alpha-level of 0.05.This difference corresponds to a mean daily improvement of 1.67 points on the EXACT symptom score; Test type: Superiority or Other; p = 0.759, ANOVA — AAC were compared between treatments using an analysis of variance model adjusting for treatment and region as factors and including the baseline score as a covariate; Least sqaure mean difference = 23.7, 95% CI 2-sided [-128.3 to 175.7]

2. Secondary Outcome: Change From Baseline in COPD Assessment Tool (CAT) Score
Description: The secondary objective is to evaluate the treatment effect of once daily administrations of AQX-1125 compared to placebo over 12 weeks on the COPD Assessment Tool (CAT) score.The CAT questionnaire measures the impact of COPD on wellbeing and daily life. Participants answer 8 questions on a scale from 0 (best) to 5 (worst). The total score ranges from 0 to 40 with higher scores indicating more impact. A negative change from baseline indicates improvement. The change in total CAT score from Day 1, before taking study drug (baseline), to end of the 12 week treatment period was compared between the two treatments using an ANOVA model adjusting for treatment and region and including the baseline score as a covariate.
Time Frame: 12 weeks
Population: Full analysis set. Missing post-treatment data imputed using the last observation carried forward principle.
Measure: Least Squares Mean (95% Confidence Interval); unit: COPD Assessment Tool Score
Groups:
- AQX-1125 (200 mg): 1 x AQX-1125 capsule daily
Arm/Group | AQX-1125 (200 mg) | Placebo
Number analyzed (Participants) | 179 | 182
COPD Assessment Tool Score | -4.05 [-5.06 to -3.04] | -3.71 [-4.71 to -2.71]
Statistical Analysis 1: Comparison: AQX-1125 (200 mg) vs Placebo; ANOVA model with fixed factors treatment, region and baseline total CAT score as covariate were used. Missing post-treatment data were imputed using the Last Observation Carried Forward principle; Test type: Superiority or Other; p = 0.588, ANOVA; Least sqaure mean difference = -0.34, 95% CI 2-sided [-1.57 to 0.89]

3. Secondary Outcome: Analysis of the Number of COPD Exacerbations (Medically Treated Event (MTE))
Description: The secondary objective is to evaluate the treatment effect of once daily administrations of AQX-1125 compared to placebo over 12 weeks on the number of COPD exacerbations (MTE).
  COPD exacerbations were referred to as Medically Treated Exacerbations (MTEs) and identified as a change in symptoms and/or signs of COPD requiring prescription of one or both of: (1) Course of oral corticosteroids or (2) Antibiotic(s).
Time Frame: 12 weeks
Population: Full analysis set was used and analyzed using the negative binomial regression model with fixed factors treatment, region and time in study as offset. Adjusted means for treatment group shows number of exacerbations/year.
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of exacerbations/year
Arm/Group | AQX-1125 (200 mg) | Placebo
Number analyzed (Participants) | 200 | 198
Number of exacerbations/year | 1.776 [1.374 to 2.297] | 1.641 [1.261 to 2.135]
Statistical Analysis 1: Comparison: AQX-1125 (200 mg) vs Placebo; The number of subjects with at least one COPD exacerbation were summarised by treatment group; Test type: Superiority or Other; p = 0.646, Negative binomial regression model; Negative binomial regression model with fixed factors treatment, region and time in study as offset; Least sqaure mean difference = 1.083, 95% CI 2-sided [0.771 to 1.520]

4. Secondary Outcome: Time to First COPD Exacerbation
Description: The secondary objective is to evaluate the treatment effect of once daily administrations of AQX-1125 compared to placebo over 12 weeks on the time to first exacerbation requiring medical intervention of oral corticosteroids and/or antibiotics.
Time Frame: 12 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: day(s)
Arm/Group | AQX-1125 (200 mg) | Placebo
Number analyzed (Participants) | 200 | 198
day(s) | 38.1 (21.3) | 43.9 (24.1)

5. Secondary Outcome: The Number of Subjects With at Least One COPD Exacerbation.
Description: The number of subjects that presented with a COPD exacerbation during the 12 week treatment period.
Time Frame: 12 weeks
Population: Full analysis set.
Measure: Number; unit: participants
Arm/Group | AQX-1125 (200 mg) | Placebo
Number analyzed (Participants) | 200 | 198
participants | 48 | 51

6. Secondary Outcome: Change From Baseline in FEV1
Description: The secondary objective is to evaluate the treatment effect of once daily administrations of AQX-1125 compared to placebo over 12 weeks on forced expiratory volume in 1 second [FEV1].
  FEV1 was determined from post-bronchodilator spirometry testing done at clinic visits.
Time Frame: 12 weeks
Population: Full analysis set. Missing post-treatment data imputed using the last observation carried forward principle.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | AQX-1125 (200mg) | Placebo
Number analyzed (Participants) | 184 | 185
Liter | -0.02 [-0.06 to 0.02] | 0.01 [-0.03 to 0.06]
Statistical Analysis 1: Comparison: AQX-1125 (200mg) vs Placebo; Missing post-treatment data was imputed using the Last Observation Carried Forward principle; Test type: Superiority or Other; p = 0.226, ANOVA

7. Secondary Outcome: AQX-1125 Concentrations in Plasma (Trough Values)
Description: The secondary objectives are to evaluate the pharmacokinetics (PK) of AQX-1125 in plasma.
Time Frame: 12 weeks
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per Liter
Groups:
- AQX-1125 Week 2: AQX-1125 Week 2 PK
- AQX-1125 Week 4: AQX-1125 Week 4 PK
- AQX-1125 Week 12: Week 12 PK Week 12 PK
Arm/Group | AQX-1125 Week 2 | AQX-1125 Week 4 | AQX-1125 Week 12
Number analyzed (Participants) | 168 | 163 | 145
micrograms per Liter | 170.1 (70.5) | 163.9 (74.5) | 120.5 (80.0)

ADVERSE EVENTS:
Time Frame: 12 weeks treatment; up to 6 months safety follow-up.
Description: SAEs listed occurred in >1 subjects per treatment arm.
Arm/Group | AQX-1125 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/200 | 1/200
Serious Adverse Events (participants affected / at risk) | 6/200 | 12/200
Other Adverse Events (participants affected / at risk) | 21/200 | 21/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AQX-1125 (N=200) | Placebo (N=200)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (9) — COPD exacerbations occurring during the study should not have been reported as SAEs (as per protocol). However, 10 events were reported (1 in AQX-1125 group and 9 in placebo).
Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AQX-1125 (N=200) | Placebo (N=200)
Diarrhoea (Gastrointestinal disorders) | 11 (13) | 9 (9)
Headache (Nervous system disorders) | 12 (12) | 13 (14)

LIMITATIONS AND CAVEATS:
Secondary objective of "The frequency and severity of AEs and changes in physical exam, vital signs, ophthalmic exam, laboratory tests, weight, ECG, and con meds" was monitored throughout the study, clinically significant events were reported as AEs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators shall not publish any articles or make any presentations or communications (including any written, oral or electronic manuscript, abstract, presentation or other publication) relating to the Services, Sponsor Information, Study Drug or other Material, Deliverables or other Developments, in whole or part, without the prior written consent of the Sponsor.